CLINICAL TRIAL: NCT05284929
Title: Increased Frequencies of Certain HLA Class II Alleles DRB1 and DQB1 in PV Patients Compared to Those in Healthy Donors Have Been Reported in Various Populations and Repeatedly Confirmed. Among the Russian Population, no Studies About the Association of PV and HLA Class II Genes Have Been Conducted. Thus, the Purpose of This Study Was to Investigate HLA Class II Alleles and Haplotypes in Russian Patients With Pemphigus Vulgaris.
Brief Title: Human Leukocyte Antigen Class II (DRB1 and DQB1) Alleles and Haplotypes Frequencies in Patients With Pemphigus Vulgaris Among the Russian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sechenov University (Other)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: #03-22
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Pemphigus; Bullous Pemphigoid; Stevens-Johnson Syndrome; Toxic Epidermal Necrolyses
MeSH Terms: conditions — Pemphigus; Pemphigoid, Bullous; Stevens-Johnson Syndrome | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pemphigus
  Interventions: Genetic: A single blood sample for HLA typing
- Healthy controls
  Interventions: Genetic: A single blood sample for HLA typing

INTERVENTIONS:
Genetic: A single blood sample for HLA typing — Extracting of DNA from the blood sample using PCR-reaction

SUMMARY:
Pemphigus is a rare autoimmune life-threatening blistering condition affecting skin and mucous membranes. Pemphigus belongs to a family of polygenic disorders. Several different genes encoding molecules regulate pemphigus autoimmunity. Many trials focused on HLA investigation. Increased levels of certain HLA class II alleles frequencies in pemphigus have been reported in various populations. However, they were not investigated in the Russian population.

The aim of our study is to investigate HLA class II alleles and haplotypes in Russian patients with pemphigus.

Methods

Patients and controls

We are recruiting 120 patients with pemphigus. The diagnosis was based on clinical and histopathological findings and confirmed by immunofluorescent techniques (direct and indirect immunofluorescent tests). Before sampling, written consent was obtained from each subject. A single blood sample for HLA typing was obtained from all subjects. This study has been approved by the Ethics Committee of Sechenov University, Russia. Phenotypic and allelic frequencies were compared with healthy blood donors (n=100) registered in Sechenov University blood center.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age of patients >18 years
* Confirmed diagnosis

Exclusion Criteria:

* No as pemphigus is a life-threatening condition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 120 patients with confirmed diagnosis of pemphigus will be enrolled in the study Age >18 years Sex: both females and males
  100 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2022-11-17 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
Estimation of HLA-DRB1 and HLA-DQB1 alleles frequencies in PV patients and controls | May 2017 - 2023
  The frequencies of HLA alleles will be counted directly from genotyping data, while the frequencies of haplotypes will be estimated with an expectation-maximization algorithm using the ARLEQUIN software package (version 3.11), leading to maximum-likelihood estimates of gene frequencies. To compare the differences between frequencies in the donor and patient groups the Fisher exact test will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Sechenov University, Moscow, Russia